CLINICAL TRIAL: NCT06316297
Title: A Phase I/II, Randomized, Placebo-controlled, Multi-arm, Dose-finding Study to Evaluate the Safety, Efficacy and Immunogenicity of an Acne mRNA Vaccine Candidate in Adults With Moderate to Severe Acne 18 to 45 Years of Age
Brief Title: Study to Evaluate Safety, Efficacy and Immunogenicity of Acne mRNA Vaccine in Adults With Moderate to Severe Acne
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: VBE00001; U1111-1295-3154 (Registry Identifier: ICTRP); 2025-521740-38 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: This trial will consist of a Core Study followed by an optional Long-Term Extension (LTE). The Core Study will consist of a Sentinel Cohort A, paired with a Main Cohort, evaluating the safety and efficacy of the 2-administration regimen and a Sentinel Cohort B, evaluating the safety of the 3-administration regimen. The Sentinel Cohorts will assess the safety of the dose levels and regimens in a stepwise manner.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Core Study:
  Sentinel Cohorts: modified double-blind
  * Investigators, participants, laboratory personnel will be blinded.
  * Clinical site staff preparing/administering the study vaccines will be unblinded.
  * Sponsor study staff involved in ESDRs will be unblinded at the time of the ESDR.
  Main Cohort: modified double-blind
  * Investigators, participants, laboratory personnel and Sponsor study staff will be blinded.
  * Only clinical site staff preparing/administering the study vaccines will be unblinded.
  Long-Term Extension:
  Sentinel Cohorts and Main Cohort: double-blind
  • Investigators, participants, laboratory personnel and Sponsor study staff will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sentinel Cohort A - Experimental (Experimental): Two administrations of the Acne mRNA vaccine will be injected in three increasing doses
  Interventions: Biological: Acne mRNA vaccine
- Sentinel Cohort A - Placebo (Placebo Comparator): Two administrations of placebo will be injected
  Interventions: Other: Placebo
- Sentinel Cohort B - Experimental (Experimental): Three administrations of the Acne mRNA vaccine will be injected in two increasing doses
  Interventions: Biological: Acne mRNA vaccine
- Sentinel Cohort B - Placebo (Placebo Comparator): Three administrations of placebo will be injected
  Interventions: Other: Placebo
- Main Cohort - Experimental (Experimental): Two administrations of the Acne mRNA vaccine will be injected in three increasing doses
  Interventions: Biological: Acne mRNA vaccine
- Main Cohort - Placebo (Placebo Comparator): Two administrations of placebo will be injected
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Acne mRNA vaccine — Pharmaceutical form: Liquid suspension for injection Route of administration: intramuscular
  Arms: Main Cohort - Experimental; Sentinel Cohort A - Experimental; Sentinel Cohort B - Experimental
Other: Placebo — Pharmaceutical form: Liquid solution for injection Route of administration: intramuscular
  Arms: Main Cohort - Placebo; Sentinel Cohort A - Placebo; Sentinel Cohort B - Placebo

SUMMARY:
The purpose of the trial is to evaluate the safety, efficacy and immunogenicity of up to 3 intramuscular injections of the Acne mRNA vaccine candidate at up to three dose levels in adult participants aged 18 to 45 years with moderate to severe acne.

This trial will consist of a Core Study followed by an optional Long-Term Extension (LTE). The Core Study will consist of a Sentinel Cohort A paired with a Main Cohort, evaluating the safety and efficacy of the 2-administration regimen and a Sentinel Cohort B, evaluating the safety of the 3- administration regimen. The Sentinel Cohorts will assess the safety of the dose levels and regimens in a stepwise manner. If the participants consent to the LTE, they will be followed up for an additional 30 months after the last planned visit in the Core Study, to assess the long-term effects of the vaccine.

DETAILED DESCRIPTION:
Acne vulgaris (acne) is a highly prevalent inflammatory skin disease, especially in adolescents and young adults. Acne is estimated to affect 231 million people worldwide, therefore being one of the most prevalent diseases globally. Acne is also one of the top causes of years lived with disability and nonfatal disease burden. Despite being one of the most prevalent diseases worldwide, the mainstays of acne treatment have remained largely unchanged over the past 30 years. To date there is still no safe and effective treatment that can prevent and cure this disease.

The aim of this first-in-human (FIH), Phase I/II trial is to evaluate the safety, efficacy and immunogenicity of the Acne mRNA vaccine candidate at three different dose levels in adults aged 18 to 45 years with moderate to severe acne. The results of this FIH and proof of concept study will allow selection of the vaccine dose level to be used in Phase III pivotal efficacy trial(s) and to generate preliminary data to further select the vaccine regimen.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests as judged by the investigator
* Clinical diagnosis of moderate or severe facial acne vulgaris with Investigator's Global Assessment (IGA) score of Moderate or Severe (grade 3 or grade 4 on the 5-grade IGA scale) and ≥ 25 non-inflammatory lesions (ie, open and closed comedones) and ≥ 20 inflammatory lesions (ie, papules and pustules) and ≤ 2 nodulocystic lesions (ie, nodules and cysts)

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within 6 months prior to the first study intervention administration; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the study intervention components (eg, polyethylene glycol [PEG], polysorbate); history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances; any allergic reaction (eg, anaphylaxis) after administration of mRNA coronavirus disease 2019 (COVID-19) vaccine
* Active nodulocystic acne, acne conglobate, acne fulminans, secondary acne (eg, chloracne, drug-induced acne) or other forms of acne (eg, acne mechanica)
* Use of any acne-affecting treatment without an appropriate washout period
* Receipt of any vaccine (other than the study vaccine) in the 4 weeks preceding any study intervention administration or planned receipt of any vaccine (other than the study vaccine) in the 4 weeks following any study intervention administration
* Previous vaccination against C. acnes with an investigational vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Self-reported or documented seropositivity for human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Core Study - Sentinel Cohort A and B: Number of participants with unsolicited systemic AEs | 30 minutes after each administration
  Presence of unsolicited systemic adverse events (AEs) reported
Core Study - Sentinel Cohort A and B: Number of participants with solicited injection site and systemic reactions | Up to 7 days after each administration
  Presence of solicited injection site and systemic reactions (ie, pre-listed in the participant diary [PDi] and in the case report form [CRF])
Core Study - Sentinel Cohort A and B: Number of participants with unsolicited AEs | Up to 28 days after each administration
Core Study - Sentinel Cohort A and B: Number of participants with MAAEs | Up to 6 months after each administration
  Presence of medically attended adverse events (MAAEs)
Core Study - Sentinel Cohort A and B: Number of participants with SAEs | Up to 6 months after each administration
  Presence of all serious adverse events (SAEs)
Core Study - Sentinel Cohort A and B: Number of participants with AESIs | Up to 6 months after each administration
  Presence of AEs of special interest (AESIs)
Core Study - Sentinel Cohort A and B: Number of participants with out-of-range biological test results (including shift from baseline values) | Through 7 days after administration (Day 8)
Core Study - Main Cohort: Percentage change from baseline (Day 1) in the number of inflammatory acne lesions on face | At 2 months post last administration
Core Study - Main Cohort: Percentage change from baseline (Day 1) in the number of non-inflammatory acne lesions on face | At 2 months post last administration
Long-Term Extension - Sentinel Cohort A, B and Main Cohort: Number of participants with SAEs and AESIs | Up to 38 months after first administration
  Presence of all serious adverse events (SAEs) and adverse events of special interest (AESIs)

SECONDARY OUTCOMES:
Core Study - Sentinel Cohort A, B and Main Cohort: Vaccine-antigen-specific serum antibody titers | From baseline (Day 1) to 6 months post last administration
Core Study - Main Cohort: Absolute change from baseline (Day 1) in the number of inflammatory acne lesions on face | At1 month post first administration until 6 months post last administration
Core Study - Main Cohort: Percentage change from baseline (Day 1) in the number of inflammatory acne lesions on face | At 1 month post first administration until 6 months post last administration
Core Study - Main Cohort: Absolute change from baseline (Day 1) in the number of non-inflammatory acne lesions on face | At 1 month post first administration until 6 months post last administration
Core Study - Main Cohort: Percentage change from baseline (Day 1) in the number of non-inflammatory acne lesions on face | At 1 month post first administration until 6 months post last administration
Core Study - Main Cohort: Absolute change from baseline in IGA score | At 1 month post first administration until 6 months post last administration
Core Study - Main Cohort: Number of participants with unsolicited systemic AEs | 30 minutes after each administration
  Presence of unsolicited systemic adverse events (AEs) reported
Core Study - Main Cohort: Number of participants with solicited injection site and systemic reactions | Up to 7 days after each administration
  Presence of solicited injection site and systemic reactions (ie, pre-listed in the participant diary [PDi] and in the case report form [CRF])
Core Study - Main Cohort: Number of participants with unsolicited AEs | Up to 28 days after each administration
Core Study - Main Cohort: Number of participants with MAAEs | Up to 6 months after each administration
  Presence of medically attended adverse events (MAAEs)
Core Study - Main Cohort: Number of participants with SAEs | Up to 6 months after each administration
  Presence of all serious adverse events (SAEs)
Core Study - Main Cohort: Number of participants with AESIs | Up to 6 months after each administration
  Presence of AEs of special interest (AESIs)
Core Study - Main Cohort: Number of participants with out-of-range biological test results (including shift from baseline values) | Through 7 days after administration (Day 8)

CONTACTS AND LOCATIONS:
Locations (93):
- United States (79):
  - Center for Dermatology and Plastic Surgery- Site Number : 8400111, Scottsdale, Arizona
  - Private Practice - Dr. Francisco Badar- Site Number : 8400067, Cerritos, California
  - Encino Research Center- Site Number : 8400033, Encino, California
  - Paradigm Clinical Research Centers- Site Number : 8400064, La Mesa, California
  - Sunwise Clinical Research- Site Number : 8400108, Lafayette, California
  - Chemidox Clinical Trials- Site Number : 8400075, Lancaster, California
  - Kaiser Permanente - Los Angeles Medical Center- Site Number : 8400058, Los Angeles, California
  - LA Universal Research Center- Site Number : 8400059, Los Angeles, California
  - Alliance Clinical - West Hills- Site Number : 8400131, Los Angeles, California
  - Carbon Health - North Hollywood - NoHo West- Site Number : 8400076, North Hollywood, California
  - Northridge Clinical Trials - Northridge- Site Number : 8400053, Northridge, California
  - Profound Research - Dermatologist Medical Group of North County- Site Number : 8400099, Oceanside, California
  - Cura Clinical Research - Oxnard- Site Number : 8400062, Oxnard, California
  - Amicis Research Center, LLC- Site Number : 8400110, Palmdale, California
  - Empire Clinical Research - Pomona- Site Number : 8400055, Pomona, California
  - Peninsula Research Associates- Site Number : 8400102, Rolling Hills Estates, California
  - Artemis Institute for Clinical Research, LLC- Site Number : 8400103, San Diego, California
  - California Research Foundation- Site Number : 8400095, San Diego, California
  - NorthBay Clinical Research- Site Number : 8400066, Santa Rosa, California
  - Encore Medical Research of Boynton Beach- Site Number : 8400116, Boynton Beach, Florida
  - Driven Research- Site Number : 8400135, Coral Gables, Florida
  - HealthMed Clinical Center Inc.- Site Number : 8400071, Coral Gables, Florida
  - Universal Medical Research - Coral Gables- Site Number : 8400081, Coral Gables, Florida
  - Genomics Medical Research- Site Number : 8400120, Cutler Bay, Florida
  - Direct Helpers Research Center- Site Number : 8400118, Hialeah, Florida
  - Zenith Clinical Research- Site Number : 8400127, Hollywood, Florida
  - Encore Medical Research - Hollywood- Site Number : 8400122, Hollywood, Florida
  - Universal Medical and Research Center- Site Number : 8400079, Homestead, Florida
  - Encore Research Group-Jacksonville Center for Clinical Research- Site Number : 8400006, Jacksonville, Florida
  - K2 Summit Research LLC - Site Number : 8400063, Lady Lake, Florida
  - Dr. Manuel J Hernandez Clinical Research and Associates, Inc.- Site Number : 8400106, Miami, Florida
  - SouthCoast Research Center- Site Number : 8400114, Miami, Florida
  - Advanced Medical Research Institute - Miami- Site Number : 8400100, Miami, Florida
  - Health and Life Research Institute, LLC- Site Number : 8400070, Miami, Florida
  - WellQuest Clinical- Site Number : 8400082, Miami, Florida
  - Renstar Medical Research - Ocala - Northeast 1st Avenue- Site Number : 8400021, Ocala, Florida
  - Leading Edge Dermatology- Site Number : 8400077, Plantation, Florida
  - Nuline Clinical Trial Center- Site Number : 8400060, Pompano Beach, Florida
  - D&H Tamarac Research Center- Site Number : 8400121, Tamarac, Florida
  - TrueBlue Clinical Research- Site Number : 8400016, Tampa, Florida
  - Optimum Clinical Trial Group- Site Number : 8400125, Tampa, Florida
  - CenExel FCR Tampa- Site Number : 8400130, Tampa, Florida
  - Accel Research Sites - NeuroStudies- Site Number : 8400134, Decatur, Georgia
  - MetroMed Clinical Trials- Site Number : 8400054, Chicago, Illinois
  - AMR Chicago- Site Number : 8400019, Oak Brook, Illinois
  - NorthShore University Health System - Endeavor Health Medical Group - Skokie - Woods Drive- Site Number : 8400031, Skokie, Illinois
  - Dawes Fretzin Clinical Research- Site Number : 8400022, Indianapolis, Indiana
  - Accellacare - McFarland Clinic- Site Number : 8400045, Ames, Iowa
  - The Iowa Clinic West Des Moines Campus- Site Number : 8400084, West Des Moines, Iowa
  - Equity Medical - Bowling Green- Site Number : 8400093, Bowling Green, Kentucky
  - Louisiana Dermatology Associates- Site Number : 8400043, Baton Rouge, Louisiana
  - Clinical Trials Management - Metairie- Site Number : 8400072, Metairie, Louisiana
  - DelRicht Research - New Orleans 308- Site Number : 8400013, New Orleans, Louisiana
  - Private Practice - Dr. Lawrence J. Green- Site Number : 8400024, Rockville, Maryland
  - MetroBoston Clinical Partners - Brighton- Site Number : 8400008, Brighton, Massachusetts
  - Kuchnir Dermatology & Dermatologic Surgery- Site Number : 8400096, Marlborough, Massachusetts
  - Michigan Institute of Research- Site Number : 8400092, Allen Park, Michigan
  - Vida Clinical Studies - Dearborn Heights- Site Number : 8400074, Dearborn Heights, Michigan
  - Clinical Research Institute - Minneapolis- Site Number : 8400080, Minneapolis, Minnesota
  - MediSearch Clinical Trials- Site Number : 8400035, Saint Joseph, Missouri
  - Boeson Research - Missoula- Site Number : 8400069, Missoula, Montana
  - Las Vegas Clinical Trials- Site Number : 8400056, Las Vegas, Nevada
  - Trial Management Associates - Wilmington - Floral Parkway- Site Number : 8400104, Wilmington, North Carolina
  - Lynn Institute of Oklahoma City- Site Number : 8400004, Oklahoma City, Oklahoma
  - Best Skin Research - Camp Hill- Site Number : 8400017, Camp Hill, Pennsylvania
  - Delricht Research - Mt Pleasant Dermatology- Site Number : 8400047, Mt. Pleasant, South Carolina
  - DelRicht Research - Thompson's Station- Site Number : 8400041, Smyrna, Tennessee
  - Inquest Clinical Research - Baytown - West Baker Road- Site Number : 8400115, Baytown, Texas
  - DFW Clinical Trials- Site Number : 8400057, Carrollton, Texas
  - Modern Research Associates- Site Number : 8400094, Dallas, Texas
  - Center for Clinical Studies - Houston - Binz Street- Site Number : 8400002, Houston, Texas
  - Lone Star Clinical Research - Katy- Site Number : 8400049, Katy, Texas
  - DelRicht Research - Lockhart Matter Dermatology & Aesthetic Center- Site Number : 8400046, Prosper, Texas
  - Cope Family Medicine - Ogden Clinic- Site Number : 8400112, Bountiful, Utah
  - Alpine Research Association- Site Number : 8400050, Layton, Utah
  - CenExel JRB - Salth Lake City- Site Number : 8400128, Salt Lake City, Utah
  - Springville Dermatology - Springville- Site Number : 8400113, Springville, Utah
  - The Education & Research Foundation- Site Number : 8400036, Lynchburg, Virginia
  - Seattle Clinical Research Center- Site Number : 8400038, Seattle, Washington
- Australia (8):
  - Investigational Site Number : 0360001, Phillip, Australian Capital Territory
  - Investigational Site Number : 0360008, Kotara, New South Wales
  - Investigational Site Number : 0360003, Sydney, New South Wales
  - Investigational Site Number : 0360006, Waitara, New South Wales
  - Investigational Site Number : 0360005, Woolloongabba, Queensland
  - Investigational Site Number : 0360007, Carlton, Victoria
  - Investigational Site Number : 0360002, Melbourne, Victoria
  - Investigational Site Number : 0360009, Melbourne, Victoria
- Canada (6):
  - Investigational Site Number : 1240006, Edmonton, Alberta
  - Investigational Site Number : 1240001, Barrie, Ontario
  - Investigational Site Number : 1240004, Toronto, Ontario
  - Investigational Site Number : 1240009, Montreal, Quebec
  - Investigational Site Number : 1240007, Québec, Quebec
  - Investigational Site Number : 1240008, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VBE00001 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25729&tenant=MT_SNY_9011